CLINICAL TRIAL: NCT04172376
Title: Stereotactic Operation Integrating With Thrombolysis in Basal Ganglion Hemorrhage Evacuation II (SOITBE II)
Brief Title: Stereotactic Operation Integrating With Thrombolysis in Basal Ganglion Hemorrhage Evacuation II
Acronym: SOITBE II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Huashan Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Southern Medical University, China (Other); China-Japan Friendship Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); The Affiliated Hospital Of Southwest Medical University (Other); Tibet Autonomous Region People's Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); General Hospital of Ningxia Medical University (Other); Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-330
Record Dates: First submitted 2019-10-21; First posted 2019-11-21 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Basal Ganglia Hemorrhage
Keywords: basal ganglion hemorrhage; stereotactic surgery; thrombolysis
MeSH Terms: conditions — Basal Ganglia Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive puncture aspiration plus rt-PA (Experimental)
  Interventions: Procedure: Minimally invasive puncture aspiration plus rt-PA
- Conservative medical treatment (Active Comparator)
  Interventions: Drug: Conservative medical treatment

INTERVENTIONS:
Procedure: Minimally invasive puncture aspiration plus rt-PA — Stereotactic puncture aspiration to evacuate basal ganglion hematoma with use of thrombolytic agent
  Arms: Minimally invasive puncture aspiration plus rt-PA
Drug: Conservative medical treatment — Drugs for symptomatic treatment such as hemostasis and nerve nourishing.
  Arms: Conservative medical treatment

SUMMARY:
Spontaneous cerebral hemorrhage is one of the main causes of death and disability all over the world, accounting for 20%-30% of all cerebrovascular diseases. Minimally invasive surgery of cerebral hemorrhage, especially puncture aspiration, can improve early and long-term neurological recovery in patients with cerebral hemorrhage. Until now, no standardized practice for minimally invasive surgery of spontaneous cerebral hemorrhage has been established. Hematoma puncture and drainage based on CT scans without precise localization and personalized approach design, which may lead to poor efficacy and high risk of complications. The investigators' hospital has much experience in treating cerebral hemorrhage with stereotactic puncture and aspiration. So the investigators conduct a prospective multicenter randomized controlled clinical trial across the country to determine the therapeutic effects of puncture aspiration plus thrombolysis treatment for the perioperative and long-term recovery of patients with small hematoma in deep basal ganglia via computerized precision coordinates and personalized approach design.

DETAILED DESCRIPTION:
1. Prospective enrollment of patients with small spontaneous basal ganglia hematoma according to the inclusion and exclusion criteria in 14 major neurosurgical centers across the country to establish a multi-center clinical database of spontaneous small basal ganglia hematoma with data maintenance and update.
2. Random allocation of the patients enrolled into control group (conservative treatment with conventional drugs) or intervention group (minimally invasive puncture aspiration plus rt-PA); long-term follow-up for 6 months to compare the recent and long-term mortality rate, disability rate and related complications of the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of spontaneous basal ganglia hemorrhage by imaging (CT, CTA, etc.) with a volume of 15-30 mL calculated by ABC/2 formula and Glasgow Coma Scale score of at least 9.
2. With dysfunctions such as hematoma-related motor aphasia, sensory aphasia, hemiplegic limb muscle strength ≤ grade 3 or NIHSS score ≥ 15.
3. Hematoma volume increase <5 ml by ABC/2 formula shown by an additional CT scan after at least 6 hours of the diagnostic CT.
4. Diagnostic CT scans should be obtained within 24 hours after the onset of symptoms. Cases with unclear onset time should be excluded.
5. Randomization within 72 hours after diagnostic CT.
6. Surgery performed within 72 hours after onset.
7. SBP <180 mmHg recorded for 6 hours prior to randomization.
8. Age between 18-70 years old.
9. mRS score ≤ 1 in past medical history.
10. Patients are suitable and willing to be randomized to puncture aspiration plus rt-PA or conventional drug treatment.

Exclusion Criteria:

1. Hematoma involves thalamus, midbrain and other structures.
2. Mass effect or hydrocephalus due to intraventricular hemorrhage.
3. Imaging-based diagnosis of cerebrovascular abnormalities such as ruptured aneurysm, arteriovenous malformation (AVM) and moyamoya disease, hemorrhagic transformation of ischemic infarct and recent recurrence (within 1 year) of cerebral hemorrhage.
4. Manifestation of early stage cerebral herniation such as ipsilateral pupil changes and midline shift exceeding 1 cm.
5. Patients with unstable hematoma or with progression to intracranial hypertension syndrome.
6. Patients with any irreversible coagulopathy or known coagulation disorders; platelet count < 100,000; INR > 1.4.
7. Patients requiring long-term use of anticoagulants.
8. Patients taking dabigatran, apixaban, and/or rivaroxaban (or similar drugs of the same category) before symptoms arise.
9. Bleeding in other sites, including retroperitoneal, gastrointestinal, genitourinary or respiratory tract bleeding; superficial or skin surface bleeding, mainly in the vascular puncture sites or transvenous approaches (e.g. arterial puncture, venous incision, etc.), or the recent surgical sites.
10. Patients who may be pregnant in the near future or are already pregnant.
11. Patients previously enrolled in this study.
12. Patients participating in other interventional medical research or clinical trials at the same time. Patients enrolled in observational, natural history and/or epidemiological studies (without intervention) are eligible for this trial.
13. Patients with an expected survival of less than 6 months.
14. Patients with severe co-morbidity (including hepatic, renal, gastrointestinal, respiratory, cardiovascular, endocrine, immune and/or hematological disorders) which would affect the outcome assessment.
15. Patients with mechanical heart valve. Biological valves are acceptable.
16. Patients with risk of embolism (including a history of left heart thrombus, mitral stenosis with atrial fibrillation, acute pericarditis or subacute bacterial endocarditis). Atrial fibrillation without mitral stenosis is acceptable.
17. Patients with co-morbidities that would be detrimental if the study begins according to investigators.
18. Lost to follow-up or poor compliance due to various reasons (such as geographical and social factors, drug or alcohol abuse, etc.)
19. Patient or his or her legal guardian/representative is unable or unwilling to give the written informed consent.
20. Patients is in a condition that is not suitable for puncture aspiration plus rt-PA treatment.

Early termination criteria:

1. Serious adverse events related to minimally invasive treatment
2. Interim analysis shows a significant difference in efficacy between the conservative and surgical groups.

Dropout criteria:

Patients who cannot be followed up during the study period are considered dropout. Dropout patients are followed up by telephone, mail or outpatient visits and the reason for the dropout and the last follow-up information should be collected as much as possible.

Elimination criteria:

Patients whose disease-related biological or imaging data are not retained should be discussed for elimination by investigators and statisticians before final analysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of ADL score | at 6 months of follow-up
  ADL: Activities of Daily Living, ranges from 0-100, a higher ADL score means a better situation.

SECONDARY OUTCOMES:
Hematoma clearance rate | at 1 day and 1 month after treatment
Change in GCS score | at 1 month after treatment
  GCS: Glasgow Coma Scale, ranges from 3-15, a higher GCS score means a better situation.
Mortality rate | at 6 months of follow-up
Improvement of the muscle strength of the hemiplegic limbs and aphasia | after 6 months of follow-up
Change in GCS score | at 6 months after treatment
  GCS: Glasgow Coma Scale, ranges from 3-15, a higher GCS score means a better situation.
Length of hospital stay | at 6 months after treatment
All costs of the hospital stay | at 6 months after treatment

REFERENCES:
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Background] Chiu CD, Chen CC, Shen CC, Chin LT, Ma HI, Chuang HY, Cho DY, Chu CH, Chang C. Hyperglycemia exacerbates intracerebral hemorrhage via the downregulation of aquaporin-4: temporal assessment with magnetic resonance imaging. Stroke. 2013 Jun;44(6):1682-9. doi: 10.1161/STROKEAHA.113.675983. Epub 2013 Apr 16. PMID 23592763
- [Background] Rincon F, Mayer SA. Novel therapies for intracerebral hemorrhage. Curr Opin Crit Care. 2004 Apr;10(2):94-100. doi: 10.1097/00075198-200404000-00003. PMID 15075717
- [Background] van Asch CJ, Luitse MJ, Rinkel GJ, van der Tweel I, Algra A, Klijn CJ. Incidence, case fatality, and functional outcome of intracerebral haemorrhage over time, according to age, sex, and ethnic origin: a systematic review and meta-analysis. Lancet Neurol. 2010 Feb;9(2):167-76. doi: 10.1016/S1474-4422(09)70340-0. Epub 2010 Jan 5. PMID 20056489
- [Background] Wang W, Jiang B, Sun H, Ru X, Sun D, Wang L, Wang L, Jiang Y, Li Y, Wang Y, Chen Z, Wu S, Zhang Y, Wang D, Wang Y, Feigin VL; NESS-China Investigators. Prevalence, Incidence, and Mortality of Stroke in China: Results from a Nationwide Population-Based Survey of 480 687 Adults. Circulation. 2017 Feb 21;135(8):759-771. doi: 10.1161/CIRCULATIONAHA.116.025250. Epub 2017 Jan 4. PMID 28052979
- [Background] Mayer SA, Rincon F. Treatment of intracerebral haemorrhage. Lancet Neurol. 2005 Oct;4(10):662-72. doi: 10.1016/S1474-4422(05)70195-2. PMID 16168935
- [Background] Talacchi A, Ricci UM, Caramia G, Massimo G. Basal ganglia haemorrhages: efficacy and limits of different surgical strategies. Br J Neurosurg. 2011 Apr;25(2):235-42. doi: 10.3109/02688697.2010.534203. Epub 2010 Dec 15. PMID 21158512
- [Background] Mendelow AD, Gregson BA, Fernandes HM, Murray GD, Teasdale GM, Hope DT, Karimi A, Shaw MD, Barer DH; STICH investigators. Early surgery versus initial conservative treatment in patients with spontaneous supratentorial intracerebral haematomas in the International Surgical Trial in Intracerebral Haemorrhage (STICH): a randomised trial. Lancet. 2005 Jan 29-Feb 4;365(9457):387-97. doi: 10.1016/S0140-6736(05)17826-X. PMID 15680453
- [Background] Mendelow AD, Gregson BA, Rowan EN, Murray GD, Gholkar A, Mitchell PM; STICH II Investigators. Early surgery versus initial conservative treatment in patients with spontaneous supratentorial lobar intracerebral haematomas (STICH II): a randomised trial. Lancet. 2013 Aug 3;382(9890):397-408. doi: 10.1016/S0140-6736(13)60986-1. Epub 2013 May 29. PMID 23726393
- [Background] Choo YS, Chung J, Joo JY, Kim YB, Hong CK. Borderline basal ganglia hemorrhage volume: patient selection for good clinical outcome after stereotactic catheter drainage. J Neurosurg. 2016 Nov;125(5):1242-1248. doi: 10.3171/2015.10.JNS151643. Epub 2016 Feb 12. PMID 26871205
- [Background] Wang WZ, Jiang B, Liu HM, Li D, Lu CZ, Zhao YD, Sander JW. Minimally invasive craniopuncture therapy vs. conservative treatment for spontaneous intracerebral hemorrhage: results from a randomized clinical trial in China. Int J Stroke. 2009 Feb;4(1):11-6. doi: 10.1111/j.1747-4949.2009.00239.x. PMID 19236490
- [Background] Hanley DF, Thompson RE, Muschelli J, Rosenblum M, McBee N, Lane K, Bistran-Hall AJ, Mayo SW, Keyl P, Gandhi D, Morgan TC, Ullman N, Mould WA, Carhuapoma JR, Kase C, Ziai W, Thompson CB, Yenokyan G, Huang E, Broaddus WC, Graham RS, Aldrich EF, Dodd R, Wijman C, Caron JL, Huang J, Camarata P, Mendelow AD, Gregson B, Janis S, Vespa P, Martin N, Awad I, Zuccarello M; MISTIE Investigators. Safety and efficacy of minimally invasive surgery plus alteplase in intracerebral haemorrhage evacuation (MISTIE): a randomised, controlled, open-label, phase 2 trial. Lancet Neurol. 2016 Nov;15(12):1228-1237. doi: 10.1016/S1474-4422(16)30234-4. Epub 2016 Oct 11. PMID 27751554
- [Background] Mould WA, Carhuapoma JR, Muschelli J, Lane K, Morgan TC, McBee NA, Bistran-Hall AJ, Ullman NL, Vespa P, Martin NA, Awad I, Zuccarello M, Hanley DF; MISTIE Investigators. Minimally invasive surgery plus recombinant tissue-type plasminogen activator for intracerebral hemorrhage evacuation decreases perihematomal edema. Stroke. 2013 Mar;44(3):627-34. doi: 10.1161/STROKEAHA.111.000411. Epub 2013 Feb 7. PMID 23391763
- [Background] Hanley DF, Thompson RE, Rosenblum M, Yenokyan G, Lane K, McBee N, Mayo SW, Bistran-Hall AJ, Gandhi D, Mould WA, Ullman N, Ali H, Carhuapoma JR, Kase CS, Lees KR, Dawson J, Wilson A, Betz JF, Sugar EA, Hao Y, Avadhani R, Caron JL, Harrigan MR, Carlson AP, Bulters D, LeDoux D, Huang J, Cobb C, Gupta G, Kitagawa R, Chicoine MR, Patel H, Dodd R, Camarata PJ, Wolfe S, Stadnik A, Money PL, Mitchell P, Sarabia R, Harnof S, Barzo P, Unterberg A, Teitelbaum JS, Wang W, Anderson CS, Mendelow AD, Gregson B, Janis S, Vespa P, Ziai W, Zuccarello M, Awad IA; MISTIE III Investigators. Efficacy and safety of minimally invasive surgery with thrombolysis in intracerebral haemorrhage evacuation (MISTIE III): a randomised, controlled, open-label, blinded endpoint phase 3 trial. Lancet. 2019 Mar 9;393(10175):1021-1032. doi: 10.1016/S0140-6736(19)30195-3. Epub 2019 Feb 7. PMID 30739747
- [Background] Kim YZ, Kim KH. Even in patients with a small hemorrhagic volume, stereotactic-guided evacuation of spontaneous intracerebral hemorrhage improves functional outcome. J Korean Neurosurg Soc. 2009 Aug;46(2):109-15. doi: 10.3340/jkns.2009.46.2.109. Epub 2009 Aug 31. PMID 19763212